CLINICAL TRIAL: NCT02504762
Title: HYbrid CoronAry Revascularization in DiabeticS: A Randomized Controlled Trial (Pilot)
Brief Title: HYbrid CoronAry Revascularization in DiabeticS
Acronym: HYCARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Marc Ruel MD MPH FRCSC, Cardiac Surgeon, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150338
Record Dates: First submitted 2015-06-29; First posted 2015-07-22 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Diabetes; Heart Disease
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment: HCR (Experimental): Participants will be randomized into the treatment or control group. In the treatment group, participants will be treated with PCI and MICS CABG. In the control group, participants will be treated with conventional CABG for their multivessel CAD.
  Interventions: Procedure: Treatment
- Control: Conventional CABG (Active Comparator): Participants will be randomized into the treatment or control group. In the treatment group, participants will be treated with PCI and MICS CABG. In the control group, participants will be treated with conventional CABG for their multivessel CAD.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Treatment — Hybrid Coronary Intervention = MICS CABG + Percutaneous Coronary Intervention. This study is a surgical intervention, which does not involve a drug or device intervention.
  Arms: Treatment: HCR
Procedure: Control — Conventional CABG. This study is a surgical intervention, which does not involve a drug or device intervention.
  Arms: Control: Conventional CABG

SUMMARY:
To evaluate whether an HCR strategy is more or less effective than conventional coronary artery bypass grafting (cCABG), in diabetic patients with multivessel CAD involving the left anterior descending artery (LAD), who do not present in the context of acute ST-elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
Globally, diabetes mellitus has become a major threat to human health. An increase in the prevalence of diabetes has been observed, which in part can be attributed to the aging of the population, as well as to an increase in the rate of obesity and sedentary lifestyle in Canada and the United States.1 Diabetes mellitus is an emerging epidemic with an estimate, currently, of almost 18 million confirmed cases and another 20 million patients with impaired glucose tolerance at risk to diabetes, in the United States alone.2,3

Diabetes mellitus, either Type-I or Type-II, is a very strong risk factor for the development of coronary artery disease (CAD) and stroke. Eighty percent of all deaths among diabetic patients are due to atherosclerosis, compared to about 30% among non-diabetic patients.2 A large NIH cohort study, the First National Health and Nutrition Examination Survey, revealed that heart disease mortality in the general population is declining at a much greater rate than in diabetic patients. In fact, diabetic women suffered an increase in heart disease mortality over the same time period.4,5 Furthermore, despite recent reductions in cardiovascular events amongst adults with diabetes, the absolute risk of cardiovascular events remains 2- fold greater than amongst non-diabetic individuals.6

There are various methods by which we can treat multivessel CAD in diabetic patients. Although conventional bypass (cCABG) is more beneficial than percutaneous coronary intervention (PCI) with drug eluting stents (DES) for myocardial revascularization in diabetics with multivessel CAD, diabetics are also the patients who experience the most complications, infections, and highest costs with cCABG through a sternotomy. Recently, we developed and diffused MICS CABG, which can be combined with PCI/DES to vessels other than the one at the front of the heart in order to constitute hybrid coronary revascularization (HCR). The safety and efficacy of MICS CABG was recently validated in a multicentre study from our research team, with 100% patency of the left internal thoracic artery (LITA)-LAD axis on angiography7. Potential advantages of an HCR approach in diabetics include the avoidance of a sternotomy and the potential for earlier recovery, less bleeding and transfusions, fewer infections, decreased costs, increased patient acceptance, while potentially maintaining the benefits of cCABG due to the LITA-LAD axis in a diabetic population.

Despite HCR's theoretical advantages as outlined above, it is a novel innovative approach that has not been studied in a randomized setting, nor in the context of diabetic patients. Its rationale and main research question stem from MICS CABG work by the principal investigator, as well as his recent, collaborative Lancet meta-analysis which revealed that diabetic patients with multivessel coronary disease (CAD) have better much survival with bypass surgery than with stents8. However, diabetics are also the patients who experience the most complications and infections from cCABG with incision of the breastbone. The investigators main hypothesis is therefore that a HCR strategy in diabetics with multivessel CAD will combine the benefits of bypass surgery on the artery at the front of the heart (the LAD), nearly eliminate the risk of complications and wound infection, and allow for faster recovery and improved quality of life when compared to cCABG. Other blockages would be treated with a PCI/DES to reduce the invasiveness of the procedure.

Overall, the investigators believe that the equipoise as to whether HCR is better than cCABG in diabetic patients with multivessel CAD constitutes the next important question in the diabetes/CAD field. The investigators propose to evaluate the feasibility of a definitive trial examining this question by conducting the present pilot trial.

Upon study approval, the time frame will be one year of recruitment, followed by 1 year of follow-up. Since this is a pilot trial, the investigators are assessing the feasibility of conducting this trial on diabetic patients with multivessel coronary artery disease. Should this trial be feasible, the investigators will extend the study to a full-scale study. At that time, an application will be submitted to conduct the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, aged 18 years or older;
2. Diabetes Mellitus (Type 1 or Type 2) undergoing treatment;
3. Multivessel disease involving the LAD + at least one other coronary territory (stenosis ≥ 70% in a 1.5 mm artery) in a patient referred for cCABG;
4. Angiographic lesion characteristics amenable to both PCI/DES and MICS CABG;
5. Indication for revascularization based upon objective ischemia.

Exclusion Criteria:

1. Severe congestive heart failure (class III or IV NYHA) at enrollment;
2. Left ventricular ejection fraction less than 20%;
3. Prior CABG surgery;
4. Prior heart valve surgery;
5. Prior PCI within the previous 6 months;
6. Previous tuberculosis or trauma to the chest that may have caused adhesions or LITA damage;
7. Previous stroke within 6 months or patients with stroke at more than 6 months with significant residual neurologic involvement, as reflected by a Rankin Score > 1;
8. Prior history of significant bleeding that might be expected to recur with MICS CABG or PCI/DES related anticoagulation;
9. STEMI or Q-wave MI within 72 hours prior to enrollment;
10. Planned simultaneous surgical procedure unrelated to coronary revascularization (e.g. valve repair/replacement, aneurysmectomy, carotid endarterectomy or carotid stenting);
11. Contraindication to either cCABG, MICS CABG, or PCI/DES because of a coexisting clinical condition;
12. Significant leukopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis;
13. Intolerance or contraindication to aspirin or both clopidogrel and ticagrelor;
14. Dementia with a Mini Mental Status Examination (MMSE) score of < 20;
15. Extra-cardiac illness that is expected to limit survival to less than 5 years;
16. Suspected pregnancy. A pregnancy test (urine or serum) will be administered to all women not clearly menopausal;
17. Concurrent enrollment in another clinical trial;
18. Geographic inaccessibility for the follow-up visits required by protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Assessing conventional CABG vs HCR in diabetic patients with multivessel CAD | Up to 24 months
  To determine whether a hybrid strategy to treat multivessel CAD in diabetics is more or less effective than conventional CABG

SECONDARY OUTCOMES:
≥ 95% participant adherence | Up to 24 months
  Adherence defined as ≥ 95% of the prescribed randomized revascularization index
Minimizing procedural crossovers | Up to 24 months
  Minimization of procedural crossovers in regards to patients crossing from one modality to the other, prior, during, or early failure of the planned, assigned index procedure
≥ 95% follow-up rate | Up to 24 months
  One year follow-up rates will be ≥ 95%
Number of patients we can enroll in 1 year | Up to 24 months
  How many eligible and consenting patients can be successfully enrolled in 1 year, and followed-up for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ruel, MD. MPH, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- Division of Cardiac Surgery, University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Findings from this study will be presented at conferences.

REFERENCES:
- [Background] Harris MI, Flegal KM, Cowie CC, Eberhardt MS, Goldstein DE, Little RR, Wiedmeyer HM, Byrd-Holt DD. Prevalence of diabetes, impaired fasting glucose, and impaired glucose tolerance in U.S. adults. The Third National Health and Nutrition Examination Survey, 1988-1994. Diabetes Care. 1998 Apr;21(4):518-24. doi: 10.2337/diacare.21.4.518. PMID 9571335
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of overweight and obesity among adults with diagnosed diabetes--United States, 1988-1994 and 1999-2002. MMWR Morb Mortal Wkly Rep. 2004 Nov 19;53(45):1066-8. PMID 15549021
- [Background] Grundy SM, Benjamin IJ, Burke GL, Chait A, Eckel RH, Howard BV, Mitch W, Smith SC Jr, Sowers JR. Diabetes and cardiovascular disease: a statement for healthcare professionals from the American Heart Association. Circulation. 1999 Sep 7;100(10):1134-46. doi: 10.1161/01.cir.100.10.1134. No abstract available. PMID 10477542
- [Background] Gu K, Cowie CC, Harris MI. Diabetes and decline in heart disease mortality in US adults. JAMA. 1999 Apr 14;281(14):1291-7. doi: 10.1001/jama.281.14.1291. PMID 10208144
- [Background] Kawate R, Yamakido M, Nishimoto Y, Bennett PH, Hamman RF, Knowler WC. Diabetes mellitus and its vascular complications in Japanese migrants on the Island of Hawaii. Diabetes Care. 1979 Mar-Apr;2(2):161-70. doi: 10.2337/diacare.2.2.161. PMID 520120
- [Background] Fox CS, Coady S, Sorlie PD, Levy D, Meigs JB, D'Agostino RB Sr, Wilson PW, Savage PJ. Trends in cardiovascular complications of diabetes. JAMA. 2004 Nov 24;292(20):2495-9. doi: 10.1001/jama.292.20.2495. PMID 15562129
- [Background] Ruel M, Shariff MA, Lapierre H, Goyal N, Dennie C, Sadel SM, Sohmer B, McGinn JT Jr. Results of the Minimally Invasive Coronary Artery Bypass Grafting Angiographic Patency Study. J Thorac Cardiovasc Surg. 2014 Jan;147(1):203-8. doi: 10.1016/j.jtcvs.2013.09.016. Epub 2013 Oct 30. PMID 24183338
- [Background] Verma S, Farkouh ME, Yanagawa B, Fitchett DH, Ahsan MR, Ruel M, Sud S, Gupta M, Singh S, Gupta N, Cheema AN, Leiter LA, Fedak PW, Teoh H, Latter DA, Fuster V, Friedrich JO. Comparison of coronary artery bypass surgery and percutaneous coronary intervention in patients with diabetes: a meta-analysis of randomised controlled trials. Lancet Diabetes Endocrinol. 2013 Dec;1(4):317-28. doi: 10.1016/S2213-8587(13)70089-5. Epub 2013 Sep 13. PMID 24622417
- [Background] Farkouh ME, Domanski M, Sleeper LA, Siami FS, Dangas G, Mack M, Yang M, Cohen DJ, Rosenberg Y, Solomon SD, Desai AS, Gersh BJ, Magnuson EA, Lansky A, Boineau R, Weinberger J, Ramanathan K, Sousa JE, Rankin J, Bhargava B, Buse J, Hueb W, Smith CR, Muratov V, Bansilal S, King S 3rd, Bertrand M, Fuster V; FREEDOM Trial Investigators. Strategies for multivessel revascularization in patients with diabetes. N Engl J Med. 2012 Dec 20;367(25):2375-84. doi: 10.1056/NEJMoa1211585. Epub 2012 Nov 4. PMID 23121323